CLINICAL TRIAL: NCT02288377
Title: A EUROPEAN, MULTICENTRE, PHASE II/III RANDOMISED DOUBLE-BLIND, PLACEBO CONTROLLED STUDY EVALUATING LANREOTIDE AS MAINTENANCE THERAPY IN PATIENTS WITH NON-RESECTABLE DUODENO-PANCREATIC NEUROENDOCRINE TUMOURS AFTER FIRST-LINE TREATMENT
Brief Title: A Study Evaluating Lanreotide as Maintenance Therapy in Patients With Non-Resectable Duodeno-Pancreatic Neuroendocrine Tumors (REMINET)
Acronym: REMINET
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Because of slow recruitment
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRODIGE31
Record Dates: First submitted 2014-09-23; First posted 2014-11-11 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Metastatic/Locally Advanced, Non-resectable, Duodeno-pancreatic Neuroendocrine Tumours
Keywords: Lanreotide; Duodeno-pancreatic neuroendocrine tumours; Maintenance treatment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lanreotide (Experimental): In this arm, patients will receive lanreotide 120 mg every 28 days until disease progression
  Interventions: Drug: lanreotide
- placebo (Placebo Comparator): In this arm, patients will receive placebo every 28 days until disease progression
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lanreotide — Patients will receive lanreotide 120 mg every 28 days until disease progression
  Arms: lanreotide
Drug: Placebo
  Arms: placebo

SUMMARY:
This European, prospective, multicentre, double-blind randomised study will evaluate the effect of lanreotide (120 mg every 28 days until disease progression) versus placebo in patients with metastatic/locally advanced, non-resectable, duodeno-pancreatic neuroendocrine tumours.

DETAILED DESCRIPTION:
This is a European, prospective, multicentre, double-blind randomised study evaluating lanreotide (120 mg every 28 days until disease progression) versus placebo in patients with metastatic/locally advanced, non-resectable, duodeno-pancreatic neuroendocrine tumours.

Depending on the phase II results, the study may be continued into phase III. The treatment and follow-up of patients will be the same in phase II and phase III.

After the first-line treatment, patients will be randomly assigned with a 1:1 ratio to receive either lanreotide or placebo. The study treatment should be initiated within 6 weeks following the confirmation date of stable disease or objective response.

Treatment period:

For each patient, the investigational products (lanreotide or placebo) will be provided according to a double-blind procedure until disease progression or toxicity, in accordance with the protocol.

The estimated average treatment duration for all patients is 12 months.

Follow-up period:

To evaluate overall survival, patients in phase II will have a minimum follow-up period of 12 months; if the study continues to phase III, these patients will have a maximum follow-up period of 10 years. Phase III patients will have a minimum follow-up period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic (synchronous or metachronous) or locally advanced, non-resectable, well-differentiated duodeno-pancreatic neuroendocrine tumour, of grade 1 or 2 (WHO 2010 classification; Ki-67 ≤ 20%)
* Progressive before first-line treatment
* Histologically confirmed (either on primary tumour or metastases)
* Pathological diagnosis validated by the NET consulting pathologist
* Documented stable disease or objective response after first-line treatment, within 4 weeks (28 days) prior to randomisation
* The first-line treatment will consist of either a chemotherapy or biotherapy (everolimus or sunitinib) as referred to TNCD or ENETS guidelines. Treatment must have been administered for 3 to 6 months for chemotherapy and for 6 months for biotherapy
* Non-functional tumour or gastrinoma controlled by PPIs
* Age > or = 18 years
* WHO 0, 1 or 2
* Effective contraception for male or female patients of childbearing age, defined as: oral contraceptives, intra-uterine devices, barrier contraceptive methods along with a spermicide gel, or surgical sterilisation. Female patients should use this contraception throughout the treatment period and for 6 months after the last treatment administration. Male patients should use contraception throughout the treatment period and for 3 months after the last treatment administration.
* Signed informed consent prior to initiation of any study-specific procedures or treatment.

Exclusion Criteria:

* History of haematological malignancy or other cancer, except those treated for more than 5 years and considered as cured, carcinoma in situ of the cervix and treated skin cancer (excluding melanoma)
* Poorly differentiated neuroendocrine carcinoma or NET grade 3 ENETS (Ki-67 > 20%)
* If primary resected, bone metastasis exclusively
* Pre-treatment by somatostatin long-acting analogue
* Total bilirubin ≥ 60 µmol/L
* Uncontrolled diabetes
* Contraindication to product used in the study or its components
* Tumour arising in the context of a genetic disease
* Pregnancy or lactation
* Patients unable to undergo medical follow-up due to geographical, social, psychological or legal reasons
* Concomitant participation in another clinical trial investigating a treatment during the treatment phase and within 30 days prior to the start of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Come Lepage, Pr, Principal Investigator — Federation Francophone de Cancerologie Digestive
Locations (24):
- Clinique Universitaire saint-Luc, Brussels, Belgium
- France (19):
  - CHU d'Angers - Hôtel Dieu, Angers
  - CHU - Hôpital Avicenne, Bobigny
  - CHU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU Le Bocage Service d'HGE, Dijon
  - CH Les Oudairies, La Roche-sur-Yon
  - Hôpital Edouard Herriot, Lyon
  - CHU La Timone, Marseille
  - Hôpital de la Source, Orléans
  - CHU Cochin, Paris
  - Hôpital Haut Lévêque Bat Magellan, Service d'hépato-gastroentérologie, Pessac
  - Hôpital de la Milétrie, Poitiers
  - Hôpital Robert Debré, Reims
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Hôpital Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Charite Campus Virchow Kilikum, Berlin
  - University Hospital Marburg, Marburg
- United Kingdom (2):
  - Royal Free Hospital Neuroendocrine Tumour Unit, London
  - Manchester Academic Health Sciences Centre (MAHSC), Manchester

REFERENCES:
- [Background] Lepage C, Dahan L, Bouarioua N, Toumpanakis C, Legoux JL, Le Malicot K, Guimbaud R, Smith D, Tougeron D, Lievre A, Cadiot G, Di Fiore F, Bouhier-Leporrier K, Hentic O, Faroux R, Pavel M, Borbath I, Valle JW, Rinke A, Scoazec JY, Ducreux M, Walter T. Evaluating lanreotide as maintenance therapy after first-line treatment in patients with non-resectable duodeno-pancreatic neuroendocrine tumours. Dig Liver Dis. 2017 May;49(5):568-571. doi: 10.1016/j.dld.2017.02.004. Epub 2017 Mar 11. PMID 28292641
- [Result] Guiney DG Jr, Hasegawa P, Davis CE. Homology between clindamycin resistance plasmids in Bacteroides. Plasmid. 1984 May;11(3):268-71. doi: 10.1016/0147-619x(84)90035-0. PMID 6087395
- [Derived] Lepage C, Phelip JM, Lievre A, Le-Malicot K, Dahan L, Tougeron D, Toumpanakis C, Di-Fiore F, Lombard-Bohas C, Borbath I, Coriat R, Lecomte T, Guimbaud R, Petorin C, Legoux JL, Michel P, Scoazec JY, Smith D, Walter T. Lanreotide as maintenance therapy after first-line treatment in patients with non-resectable duodeno-pancreatic neuroendocrine tumours: An international double-blind, placebo-controlled randomised phase II trial - Prodige 31 REMINET: An FFCD study. Eur J Cancer. 2022 Nov;175:31-40. doi: 10.1016/j.ejca.2022.07.033. Epub 2022 Sep 7. PMID 36087395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-three pts were randomised in 15 centres between January 2015 and October 2018.
Pre-assignment Details: The study was terminated prematurely because of slow recruitment.
Groups:
- Placebo: Patients will receive placebo every 28 days until disease progression
Period: Overall Study
Arm/Group | Placebo | Lanreotide
Started | 26 | 27
Completed | 25 | 27
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is the Intent-to-treat population, all the patients randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lanreotide | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.45) | 65.22 (10.30) | 63.25 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 13 | 15 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 1 | 1
  United Kingdom | 1 | 1 | 2
  France | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Alive and Progression-free at 6 Months
Description: The primary endpoint for this phase II study was the proportion of pts alive and progression-free at 6 months after randomisation, evaluated according to the results of the imaging assessment done by the investigator in line with RECIST 1.1 criteria.
Time Frame: 6 months
Population: 2 patients without tumor evaluation at cycle 4 nor cycle 7 were not evaluable for the primary criterion
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lanreotide
Number analyzed (Participants) | 24 | 26
Participants | 13 | 19

2. Secondary Outcome: Progression-Free Survival
Description: The progression-free survival is the time from inclusion to the first radiological progression or death (all causes). For patients alive without progression date of last news will be considered.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions compared the little sum of diameters observed durin the study (NADIR), or a measurable increase in a nontarget lesion, or the appearance of new lesions
Time Frame: up to 2 years
Population: Outcomes was evaluated on patients randomized and receiving at least one dose of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Lanreotide
Number analyzed (Participants) | 25 | 27
Months | 7.6 [3.0 to 9.0] | 19.4 [7.6 to 32.6]

3. Secondary Outcome: Overall Survival
Description: Overall survival considered all deaths, and time was calculated from randomisation to death.
Time Frame: 2 years after the end of the treatment
Population: The outcome was evaluated on randomized patients who received at least one dose of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of patients alive
Arm/Group | Placebo | Lanreotide
Number analyzed (Participants) | 25 | 27
Percentage of patients alive | 86.1 [62.1 to 95.4] | 95.0 [69.5 to 99.3]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment, on average of 24 months
Description: Toxicities were collected before each injection of treatment up to the end of the treatment each 28 days. The study treatment was given until withdrawal of the patients for any reason (Toxicities, progression or any other medical reason)
Arm/Group | Placebo | Lanreotide
All-Cause Mortality (participants affected / at risk) | 7/25 | 2/27
Serious Adverse Events (participants affected / at risk) | 3/25 | 5/27
Other Adverse Events (participants affected / at risk) | 6/25 | 9/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Lanreotide (N=27)
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholangitis and Malignant biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis and Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | Lanreotide (N=27)
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-11-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT02288377/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT02288377/SAP_001.pdf